CLINICAL TRIAL: NCT06452576
Title: Use of Vibration During Constraint-induced Movement Therapy
Acronym: CPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Na Jin Seo, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Pro00137672
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Hemiparesis
Keywords: constraint-induced movement therapy
MeSH Terms: conditions — Paresis | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wear vibrating watch during therapy (Experimental): The watch worn on the affected wrist vibrates during therapy.
  Interventions: Device: Vibration; Behavioral: constraint-induced movement therapy
- Wear non-vibrating watch during therapy (Placebo Comparator): The watch worn on the affected wrist does not vibrate during therapy.
  Interventions: Behavioral: constraint-induced movement therapy

INTERVENTIONS:
Device: Vibration — Watch vibrates.
  Arms: Wear vibrating watch during therapy
Behavioral: constraint-induced movement therapy — A splint or mitt is placed on the stronger, unaffected hand to encourage use of the affected upper limb in therapy.

SUMMARY:
The purpose of this study is to determine whether the hand function will improve more by using low-level vibration during constraint-induced movement therapy (CIMT), compared to CIMT alone without vibration.

DETAILED DESCRIPTION:
The low-level vibration has been shown to increase therapy outcome when used as an adjunct to therapy in adults with hemiparesis. Children who participates in the CIMT camp at MUSC will be recruited to take part in the study. Participating children will wear a watch device on their weaker arm during CIMT. The watch will vibrate only for the children who were assigned to the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral upper limb motor weakness
* Can use the affected upper limb as a gross assist during play and self-care activities
* Ambulatory for their age with intact balance and protective reactions in the less involved upper limb.

Exclusion Criteria:

* Developmental delays limiting spontaneous use of the affected upper limb
* Other health impairment

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Box and Block Test | pre-therapy and post-therapy, up to 5 consecutive days
  number of blocks moved in a minute

CONTACTS AND LOCATIONS:
Overall Officials: Na Jin Seo, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided